CLINICAL TRIAL: NCT04477291
Title: A Phase 1a/b Trial of CG-806 in Patients With Relapsed/Refractory Acute Myeloid Leukemia or Higher-Risk Myelodysplastic Syndromes
Brief Title: A Study of CG-806 in Patients With Relapsed or Refractory AML or Higher-Risk MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in corporate strategy
Sponsor: Aptose Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APTO-CG-806-03
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: CG-806; Aptose; FLT3; FLT3-ITD; D835Y; F691L; BTK; C481S; TP53; NRAS; IDH1; BCL2; Gilteritinib; Quizartinib; Midostaurin; Crenolanib; Venetoclax; Ibrutinib; Acalabrutinib; Zanubrutinib; LOXO-305; ARQ 531; AML; Acute Myeloid Leukemia; MDS; Myelodysplastic Syndrome; CLL; Chronic Lymphocytic Leukemia; Resistant; Refractory; Relapsed; Intolerant; Kinase Inhibitor; Non covalent; Luxeptinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Dose Escalation and Expansion; CG-806 will be given orally in ascending doses in patients with relapsed or refractory AML or higher-risk MDS (escalation cohort), until the maximum tolerated dose or candidate recommended Phase 2 dose is reached. Followed up by up to 50 patients enrolled in the expansion cohort at the recommended dose.
  Interventions: Drug: CG-806

INTERVENTIONS:
Drug: CG-806 — CG-806 will be given orally in ascending doses starting at 450 mg PO BID until the maximum tolerated dose or candidate recommended Phase 2 dose is reached.

SUMMARY:
This study is being done to evaluate the safety, tolerability and antitumor activity of oral CG-806 (luxeptinib) for the treatment of patients with Acute Myeloid Leukemia (except APML), secondary AML, therapy-related AML, or higher-risk MDS, whose disease has relapsed, is refractory or who are ineligible for or intolerant of intensive chemotherapy or transplantation.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1 a/b dose escalation study of safety, pharmacodynamics, and pharmacokinetics of CG-806 in ascending cohorts (3+3 design) to determine the MTD or recommended dose in patients with relapsed or refractory Acute Myeloid Leukemia (except APML), secondary AML, therapy-related AML, or higher-risk MDS whose disease has relapsed, is refractory or who are ineligible for or intolerant of intensive chemotherapy or transplantation. This is to be followed by a cohort expansion phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 years
* Life expectancy of at least 3 months
* ECOG Performance Status ≤ 2
* Patients must be able to swallow capsules
* Adequate hematologic parameters, unless cytopenias are disease caused
* Adequate renal, liver and cardiac functions

Key Exclusion Criteria:

* Patients with GVHD requiring systemic immunosuppressive therapy
* Uncontrolled leptomeningeal disease, auto-immune hemolytic anemia and uncontrolled and clinically significant disease related metabolic disorder
* Clinically significant leukostasis
* Treatment with other investigational drugs or receipt of cytotoxic therapy within 14 days prior to first study treatment administration
* Receipt of cellular immunotherapeutic agents within 4 weeks prior to first study treatment administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events of CG-806 | At the end of Cycle 1 (each cycle is 28 days)
  Patients will be assessed for adverse events during all cycles of treatment and for dose limiting toxicities in Cycle 1 (28-days). Dose escalation to a higher dose level will be considered if none of the first three patients who complete Cycle 1 (28-days) at a given dose level experience a dose limiting toxicity or if only 1 of 6 patients at a given dose level experience a dose-limiting toxicity.
Establish a CG-806 dose that maintains a biologically active plasma concentration | At the end of Cycle 1 (each cycle is 28 days)
  To determine the dose of CG-806 given orally every 12 hours daily that maintains a biologically active plasma concentration during 28-day cycles.
Establish a recommended dose for future development of CG-806 | At the end of Cycle 1 (each cycle is 28 days)
  To establish the maximum tolerated dose and/or recommended Phase 2 dose (RP2D) of CG-806 for future clinical trials in patients with AML and other advanced myeloid malignancies.

SECONDARY OUTCOMES:
Pharmacokinetics variables including maximum plasma concentration (Cmax). | At the end of Cycle 1 (each cycle is 28 days)
  Pharmacokinetics variables including maximum plasma concentration at various timepoints.
Pharmacokinetics variables including minimum plasma concentration (Cmin) | At the end of Cycle 1 (each cycle is 28 days)
  Pharmacokinetics variables including minimum plasma concentration at various timepoints.
Pharmacokinetics variables including area under the curve (AUC) | At the end of Cycle 1 (each cycle is 28 days)
  Pharmacokinetics variables including plasma concentration at various timepoints.
Pharmacokinetics variables including volume of distribution | At the end of Cycle 1 (each cycle is 28 days)
  Pharmacokinetics variables including plasma concentration at various timepoints.
Pharmacokinetics variables including clearance | At the end of Cycle 1 (each cycle is 28 days)
  Pharmacokinetics variables including plasma concentration at various timepoints.
Pharmacokinetics variables including plasma half-life. | At the end of Cycle 1 (each cycle is 28 days)
  Pharmacokinetics variables including plasma concentration at various timepoints.
To determine the ability of CG-806 to modulate the expression or activity of pharmacodynamic biomarkers of drug effect. | At the end of Cycle 1 (each cycle is 28 days)
  To determine the ability of CG-806 to modulate the expression or activity of pharmacodynamic biomarkers of drug effect.
To assess patients for evidence of anti-tumor activity of CG-806 based on hematologic, bone marrow, physical examination, evaluations | At the end of Cycle 1 (each cycle is 28 days)
  To assess patients for evidence of anti-tumor activity of CG-806 based on hematologic, bone marrow, physical examination, and FDG PET-CT imaging evaluations.
To determine the Relative Bioavailability of Generation 3 formulation given to up to 18 patients on Cycle 1 Day -3 compared to Generation 1 formulation of study drug given to patients during Cycle 1. | At the end of Cycle 1 (each cycle is 28 days)
  Compare G1 to G3 pharmacokinetics variables including maximum plasma concentration (Cmax)
To determine the Relative Bioavailability of Generation 3 formulation given to up to 18 patients on Cycle 1 Day -3 compared to Generation 1 formulation of study drug given to patients during Cycle 1. | At the end of Cycle 1 (each cycle is 28 days)
  Compare G1 to G3 Pharmacokinetics variables including minimum plasma concentration (Cmin)
To determine the Relative Bioavailability of Generation 3 formulation given to up to 18 patients on Cycle 1 Day -3 compared to Generation 1 formulation of study drug given to patients during Cycle 1. | At the end of Cycle 1 (each cycle is 28 days)
  Compare G1 to G3 Pharmacokinetics variables including area under the curve (AUC)
To determine the Relative Bioavailability of Generation 3 formulation given to up to 18 | At the end of Cycle 1 (each cycle is 28 days)
  Compare G1 to G3 Pharmacokinetics variables including volume of distribution
To determine the Relative Bioavailability of Generation 3 formulation given to up to 18 | At the end of Cycle 1 (each cycle is 28 days)
  Compare G1 to G3 Pharmacokinetics variables including clearance
Compare G1 to G3 Pharmacokinetics variables including clearance | At the end of Cycle 1 (each cycle is 28 days)
  Compare G1 to G3 Pharmacokinetics variables including plasma half-life.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Bejar, MD, PhD, Study Director — Aptose Biosciences Inc.
Locations (10):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Ochsner Healthcare, New Orleans, Louisiana
  - Atlantic Hematological Oncology Center, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu G, Zhang W, Basyal M, Nishida Y, Mizumo H, Ly C, Zhang H, Rice WG, Andreeff M. The multi-kinase inhibitor CG-806 exerts anti-cancer activity against acute myeloid leukemia by co-targeting FLT3, BTK, and aurora kinases. Leuk Lymphoma. 2024 Nov;65(11):1659-1674. doi: 10.1080/10428194.2024.2364839. Epub 2024 Jun 13. PMID 38871487
- [Derived] Yu G, Zhang W, Zhang H, Ly C, Basyal M, Rice WG, Andreeff M. The multi-kinase inhibitor CG-806 exerts anti-cancer activity against acute myeloid leukemia by co-targeting FLT3, BTK, and Aurora kinases. Res Sq [Preprint]. 2023 Feb 22:rs.3.rs-2570204. doi: 10.21203/rs.3.rs-2570204/v1. PMID 36865133